CLINICAL TRIAL: NCT03709433
Title: An ACT Skills Group and Mobile App for Worry
Brief Title: Open Trial of an ACT Skills Group and Mobile App for Worry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Michael Twohig, Ph.D., Professor, Utah State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9528
Record Dates: First submitted 2018-10-09; First posted 2018-10-17 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: All participants will receive the same active treatment (acceptance and commitment therapy groups and a mobile app)
Masking Description: No masking will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT groups and mobile app (Experimental): Participants will receive six two-hour weekly sessions of acceptance and commitment therapy (ACT) in a group format. They will also access the ACT Daily mobile app, which helps participants practice ACT skills in the moment, for the duration of the study (10-14 weeks depending on when the participant completes the baseline assessment.) Sessions use metaphors, experiential exercises, and discussion to target core ACT skills: acceptance, defusion, present-moment awareness, self-as-context, values, and committed action. The mobile app includes metaphors and experiential exercises to aid with all of these skills except self-as-context. Participants will be asked to use the app to practice these skills and to complete behavioral commitments linked to their values between sessions.
  Interventions: Behavioral: ACT groups and mobile app

INTERVENTIONS:
Behavioral: ACT groups and mobile app — See arm description.

SUMMARY:
This study is an open trial of acceptance and commitment therapy (ACT) groups combined with a mobile app for the treatment of Generalized Anxiety Disorder (GAD). The goal of this study is to evaluate if ACT groups and a mobile app are efficacious and acceptable in the treatment of GAD.

Study hypotheses are:

1. Group ACT will lead to improvement in worry, anxiety, comorbid depression, functioning, and well-being.
2. Group ACT will also lead to improvement in theoretically relevant processes, namely psychological inflexibility, anxiety-related fusion, mindfulness, and progress towards values.
3. Combining a mobile app with group ACT will be credible, acceptable, and satisfactory to participants.

DETAILED DESCRIPTION:
Participants and power:

Each group will include 6-12 participants. The target sample size is 36 participants, which would provide good power (0.90) to detect a medium effect size in a repeated-measures ANOVA with three time points and requires running at least 3 groups.

All clinics on the Utah State University campus will be asked to refer their waitlist clients to the group, if appropriate (e.g., client presented with significant worry). Local private practitioners in the Cache Valley, Utah area may also be notified about the option to refer their waitlist clients to the group. Fliers will be posted on the Utah State University campus and in the local community and distributed to providers to provide more information on the study. Fliers will direct interested individuals to contact the researchers. The study will also be listed on the Utah State University Contextual Behavioral Science Lab website with a link to the pre-screening.

Procedures:

Individuals who contact the researchers expressing interest will be sent more information on study procedures and asked to complete a brief online pre-screening specific to this study.

If potential participants are likely to be eligible based on the online pre-screening, they will be asked to schedule an initial assessment. They will be asked to review a consent form and given an opportunity to ask any questions. Those who decide to participate and sign the consent form will be administered the MINI International Neuropsychiatric Interview to check eligibility (i.e., GAD diagnosis, no serious mental illness), then asked to complete a series of self-report measures hosted on Qualtrics on an iPad to establish a baseline.

The group intervention will begin when the groups are filled. There will be no cost or compensation for participating in the groups. They will be facilitated by two doctoral students with training in ACT. Participants will be informed about and trained in using the ACT Daily mobile app at the first group and reminded about how to use it at each weekly group. Reminders about using the app will also be sent weekly through email or text to participants in the follow-up period.

Participants will be asked to complete a credibility questionnaire on paper at the end of the first session. They will be asked to complete an online post-treatment survey after the group sessions conclude, and a final online follow-up survey one month later.

Intervention:

The group therapy intervention consists of six weekly sessions of acceptance and commitment therapy (ACT). Each session will be two hours long. The intervention was developed based on established ACT protocols and adapted to fit the group format and generalized anxiety. The intervention uses metaphors, experiential exercises, and discussion to target the core elements of ACT: acceptance, defusion, present moment awareness, self-as-context, values, and committed action. Groups will be closed (i.e. new group members will not be added as sessions progress). Sessions will be video recorded for the purposes of training and supervision and to allow for a review of treatment fidelity.

The ACT Daily mobile app is hosted on Qualtrics and teaches a variety of ACT skills targeting acceptance, defusion, present moment awareness, values, and committed action. Users will answer some brief questions regarding their current symptoms and psychological flexibility and then be recommended a tailored skill relevant to the psychological flexibility process that they report struggling with the most in the moment.

ELIGIBILITY:
Inclusion criteria:

1. Seeking treatment for worry
2. Fluent in English
3. At least 18 years old
4. Have no serious mental illness
5. Not currently receiving other treatment
6. Meeting diagnostic criteria for generalized anxiety disorder

Exclusion criteria mirror inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Penn State Worry Questionnaire (PSWQ) | At posttreatment (6-10 weeks after baseline)
  The PSWQ is a 16-item self-report measure of problematic worry. The PSWQ has validity and reliability in clinical samples.

SECONDARY OUTCOMES:
Penn State Worry Questionnaire (PSWQ) | One month after the posttreatment survey is administered (10-14 weeks after baseline)
  The PSWQ is a 16-item self-report measure of problematic worry. The PSWQ has validity and reliability in clinical samples.
State-Trait Anxiety Inventory (STAI) - Trait Subscale | At posttreatment (6-10 weeks after baseline)
  The Trait subscale of the STAI is a 20-item self-report measure of trait anxiety. The STAI-T has demonstrated validity and reliability.
State-Trait Anxiety Inventory (STAI) - Trait Subscale | One month after the posttreatment survey is administered (10-14 weeks after baseline)
  The Trait subscale of the STAI is a 20-item self-report measure of trait anxiety. The STAI-T has demonstrated validity and reliability.
Beck Depression Inventory-II (BDI-II) | At posttreatment (6-10 weeks after baseline)
  The BDI-II is a 21-item measure of depressive symptoms. It had good reliability and validity.
Beck Depression Inventory-II (BDI-II) | One month after the posttreatment survey is administered (10-14 weeks after baseline)
  The BDI-II is a 21-item measure of depressive symptoms. It had good reliability and validity in clinical samples.
Acceptance and Action Questionnaire (AAQ-II) | At posttreatment (6-10 weeks after baseline)
  The AAQ-II is a 7-item measure of psychological inflexibility. It has demonstrated good reliability and validity.
Acceptance and Action Questionnaire (AAQ-II) | One month after the posttreatment survey is administered (10-14 weeks after baseline)
  The AAQ-II is a 7-item measure of psychological inflexibility. It has demonstrated good reliability and validity.
Believability of Anxious Thoughts and Feelings (BAFT) Questionnaire | At posttreatment (6-10 weeks after baseline)
  The BAFT is a 16-item measure of fusion with anxious thoughts and feelings. It has demonstrated reliability and validity.
Believability of Anxious Thoughts and Feelings (BAFT) Questionnaire | One month after the posttreatment survey is administered (10-14 weeks after baseline)
  The BAFT is a 16-item measure of fusion with anxious thoughts and feelings. It has demonstrated reliability and validity.
Mindful Attention Awareness Scale (MAAS) | At posttreatment (6-10 weeks after baseline)
  The MAAS is a 15-item measure of mindful awareness of one's experience. It has demonstrated reliability and validity. Each item is rated from 1 to 6, and a mean score is of all items is taken, therefore the overall score range is 1 to 6 with higher scores indicating higher mindfulness.
Mindful Attention Awareness Scale (MAAS) | One month after the posttreatment survey is administered (10-14 weeks after baseline)
  The MAAS is a 15-item measure of mindful awareness of one's experience. It has demonstrated reliability and validity. Each item is rated from 1 to 6, and a mean score is of all items is taken, therefore the overall score range is 1 to 6 with higher scores indicating higher mindfulness.
Valuing Questionnaire (VQ) - Progress subscale | At posttreatment (6-10 weeks after baseline)
  The Progress subscale of the VQ is a 5-item measure of progress toward one's personal values. It has good validity and internal consistency.
Valuing Questionnaire (VQ) - Progress subscale | One month after the posttreatment survey is administered (10-14 weeks after baseline)
  The Progress subscale of the VQ is a 5-item measure of progress toward one's personal values. It has good validity and internal consistency.
PROMIS 8a Satisfaction with Social Roles and Activities | At posttreatment (6-10 weeks after baseline)
  This scale is an 8-item measure of the degree to which one feels satisfied with their ability to participate in social roles and activities. This measure was developed through item response theory and has demonstrated good reliability and validity.
PROMIS 8a Satisfaction with Social Roles and Activities | One month after the posttreatment survey is administered (10-14 weeks after baseline)
  This scale is an 8-item measure of the degree to which one feels satisfied with their ability to participate in social roles and activities. This measure was developed through item response theory and has demonstrated good reliability and validity.
Mental Health Continuum-Short Form (MHC-SF) | At posttreatment (6-10 weeks after baseline)
  The MHC-SF is a 14-item measure of psychological and social well-being. It has shown good reliability and validity.
Mental Health Continuum-Short Form (MHC-SF) | One month after the posttreatment survey is administered (10-14 weeks after baseline)
  The MHC-SF is a 14-item measure of psychological and social well-being. It has shown good reliability and validity.
Credibility/Expectancy Questionnaire (CEQ) | At the end of the first group therapy session, 0-4 weeks after baseline
  The CEQ is a 6-item measure of the credibility of a treatment approach and expectations of treatment outcomes. This measure has good reliability.
Mobile app question: "How much are you....Feeling nervous, anxious, or on edge" | Each time participants use the mobile app (intervention and follow-up period). This time period will begin 0-4 weeks after baseline and end 10-14 weeks after baseline.
  This item was taken from the GAD-7, a well-validated measure of generalized anxiety. It will be used for an initial assessment each time participants begin to use the mobile app, and again after they practice one of the mobile app skills. It will be rated from 0-100.
Mobile app question: "How much are you....Worrying too much about different things" | Each time participants use the mobile app (intervention and follow-up period). This time period will begin 0-4 weeks after baseline and end 10-14 weeks after baseline.
  This item was taken from the GAD-7, a well-validated measure of generalized anxiety. It will be used for an initial assessment each time participants begin to use the mobile app, and again after they practice one of the mobile app skills. It will be rated from 0-100.
Mobile app question: "How much are you....Feeling down, depressed, or hopeless" | Each time participants use the mobile app (intervention and follow-up period). This time period will begin 0-4 weeks after baseline and end 10-14 weeks after baseline.
  This item was taken from the PHQ-9, a well-validated measure of depression. It will be used for an initial assessment each time participants begin to use the mobile app, and again after they practice one of the mobile app skills. It will be rated from 0-100.
Mobile app question: "How much are you....Fighting your feelings" | Each time participants use the mobile app (intervention and follow-up period). This time period will begin 0-4 weeks after baseline and end 10-14 weeks after baseline.
  This item assesses momentary experiential avoidance. It is lacking full validation but has been used successfully in previous mobile app research.
Mobile app question: "How much are you....Stuck in thoughts" | Each time participants use the mobile app (intervention and follow-up period). This time period will begin 0-4 weeks after baseline and end 10-14 weeks after baseline.
  This item assesses momentary cognitive fusion. It is lacking full validation but has been used successfully in previous mobile app research.
Mobile app question: "How much are you....Running on autopilot" | Each time participants use the mobile app (intervention and follow-up period). This time period will begin 0-4 weeks after baseline and end 10-14 weeks after baseline.
  This item assesses momentary inattention. It is lacking full validation but has been used successfully in previous mobile app research.
Mobile app question: "How much are you....Disconnected from values" | Each time participants use the mobile app (intervention and follow-up period). This time period will begin 0-4 weeks after baseline and end 10-14 weeks after baseline.
  This item assesses momentary values obstruction. It is lacking full validation but has been used successfully in previous mobile app research.
Treatment Evaluation Inventory-Short Form (TEI-SF) | At posttreatment (6-10 weeks after baseline)
  The TEI-SF is a 9-item measure of treatment acceptability. In this study two items were omitted and others were revised to be appropriate for the present sample. This measure has good reliability and has been demonstrated to discriminate between different treatments.
Novel satisfaction items | At posttreatment (6-10 weeks after baseline)
  13 novel items were developed assessing satisfaction with the intervention (both overall and for specific components).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Twohig, PhD, Principal Investigator — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fleming, J. E., & Kocovski, N. L. (2014). MINDFULNESS AND ACCEPTANCE-BASED GROUP THERAPY FOR SOCIAL ANXIETY DISORDER: A Treatment Manual (2nd ed.). Retrieved from https://contextualscience.org/mindfulness_and_acceptancebased_group_therapy_for_1
- [Background] Boone, M. S., & Cannici, J. (2013). Acceptance and commitment therapy (ACT) in groups. In Pistorello, J., (Ed.). Acceptance and mindfulness for counseling college students: Theory and practical applications for intervention, prevention, and outreach. Oakland, CA: New Harbinger.
- [Background] Twohig, M. (2004). ACT for OCD: Abbreviated Treatment Manual. (Unpublished treatment protocol). University of Nevada, Reno.
- [Background] Hayes, S. C., Strosahl, K., & Wilson, K. G. (2012). Acceptance and Commitment Therapy, Second Edition: The Process and Practice of Mindful Change. New York: Guilford Press.
- [Background] Levin, M.E., Haeger, J. & Cruz, R.A. (In Press). Tailoring acceptance and commitment therapy skill coaching in-the-moment through smartphones: Results from a randomized controlled trial. Mindfulness.
- [Background] Meyer TJ, Miller ML, Metzger RL, Borkovec TD. Development and validation of the Penn State Worry Questionnaire. Behav Res Ther. 1990;28(6):487-95. doi: 10.1016/0005-7967(90)90135-6. PMID 2076086
- [Background] Molina, S., & Borkovec, T. D. (1994). The Penn State Worry Questionnaire: Psychometric properties and associated characteristics. In G. C. L. Davey & F. Tallis (Eds.), Wiley series in clinical psychology. Worrying: Perspectives on theory, assessment and treatment (pp. 265-283). Oxford, England: John Wiley & Sons.
- [Background] Spielberger, C. D. (1983). State-Trait Anxiety Inventory (Form Y). Redwood City, CA: Mind Garden.
- [Background] Segal DL, Coolidge FL, Cahill BS, O'Riley AA. Psychometric properties of the Beck Depression Inventory II (BDI-II) among community-dwelling older adults. Behav Modif. 2008 Jan;32(1):3-20. doi: 10.1177/0145445507303833. PMID 18096969
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Herzberg KN, Sheppard SC, Forsyth JP, Crede M, Earleywine M, Eifert GH. The Believability of Anxious Feelings and Thoughts Questionnaire (BAFT): a psychometric evaluation of cognitive fusion in a nonclinical and highly anxious community sample. Psychol Assess. 2012 Dec;24(4):877-91. doi: 10.1037/a0027782. Epub 2012 Apr 9. PMID 22486595
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Smout, M., Davies, M., Burns, N., & Christie, A. (2014). Development of the valuing questionnaire (VQ). Journal of Contextual Behavioral Science, 3, 164-172.
- [Background] Hahn EA, DeWalt DA, Bode RK, Garcia SF, DeVellis RF, Correia H, Cella D; PROMIS Cooperative Group. New English and Spanish social health measures will facilitate evaluating health determinants. Health Psychol. 2014 May;33(5):490-9. doi: 10.1037/hea0000055. Epub 2014 Jan 20. PMID 24447188
- [Background] Lamers SM, Westerhof GJ, Bohlmeijer ET, ten Klooster PM, Keyes CL. Evaluating the psychometric properties of the Mental Health Continuum-Short Form (MHC-SF). J Clin Psychol. 2011 Jan;67(1):99-110. doi: 10.1002/jclp.20741. PMID 20973032
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Kelley, M. L., Heffer, R. W., Gresham, F. M., & Elliot, S. N. (1989). Development of a modified Treatment Evaluation Inventory. Journal of Psychopathology and Behavioral Assessment, 11, 235-247. doi:10.1007/BF00960495